CLINICAL TRIAL: NCT03455374
Title: Diamondback Atherectomy With OCT Visualization for Calcified PAD Lesions for Calcified Peripheral Vascular Disease Lesions
Brief Title: Diamondback in Peripheral Vascular Disease
Acronym: DIAMOND-PAD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI/Sponsor mutual agreement due to poor enrollment
Sponsor: Arkansas Heart Hospital (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20171653
Record Dates: First submitted 2018-02-08; First posted 2018-03-06 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Peripheral Vascular Diseases; Critical Limb Ischemia
MeSH Terms: conditions — Peripheral Vascular Diseases; Chronic Limb-Threatening Ischemia | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment with CSI atherectomy device (Experimental): removal of the plaque from vessel wall by optical coherence tomography
  Interventions: Device: Treatment with CSI atherectomy device

INTERVENTIONS:
Device: Treatment with CSI atherectomy device — Following peripheral angiography, patients with significant SFA or below the knee artery disease (≥ 50%) or total occlusions (100%) will have a baseline OCT imaging of the target vessel and the lesion be treated with proper size CSI burr. Repeat OCT imaging will be performed after CSI. Drug eluting balloon angioplasty may be performed in discretion of the operator. If DEB is used, a final OCT imaging will be performed to assess lesion expansion and possible dissections. Balloon sizing will be based on 1:1 vessel ratio with the length covering from minimally diseased distal segment to minimally diseased proximal segment. We will try to avoid use of stents.

SUMMARY:
This is a prospective, nonrandomized, single-arm study using CSI Orbital Atherectomy System in patients with PAD (total occlusions or significant stenosis). Patients will be enrolled if they have claudication and/or critical limb ischemia, and identifiable PAD disease with moderate to severe calcification on Computer Tomography Angiogram (PCA) or peripheral angiogram requiring percutaneous peripheral intervention (PPI).

DETAILED DESCRIPTION:
Orbital atherectomy (OA) is one of the most commonly used modalities for the treatment of obstructive femoral-popliteal PAD, especially in patients with large and calcified atherosclerotic plaques, either as stand alone or with subsequent drug-coated balloon angioplasty or stent implantation. These atherectomy procedures were primarily guided by peripheral angiography which has significant resolution limitations in regards to the plaque morphology and characteristics such as extent of calcification, and how deep the cuts are made in the vessel wall.

Optical coherence tomography (OCT) has recently emerged as a novel imaging modality. OCT imaging has been used both in coronary as well as in peripheral circulation extensively with no significant device related adverse effects. Previous research has shown the feasibility and safety of OCT use for peripheral artery imaging and its use in plaque characterization. The hypothesis for this study is that; use of diamond back atherectomy device will lead to effective removal of plaque in moderate to heavily calcified arteries without damaging deep into the adventitia or EEL or the adjacent healthy vessel wall and thus will lead to a favorable vascular response during follow up.

ELIGIBILITY:
Inclusion Criteria:

* • Patient with lower extremity claudication and PAD due to significant SFA or below the knee stenosis (50%≤99%) or total occlusions (100%) that affects the quality of life despite medical therapy.

  * Evidence of significant SFA or below the knee disease involving the most symptomatic limb by noninvasive vascular testing with the use of the following:

    * ABI: <0.9 (If ABI>1.4, SFA systolic acceleration time should be > 140 milliseconds);
    * TBI: <0.6;
    * Computed Tomographic Angiography (CTA) confirming at least a 50% SFA stenosis with moderate to severe calcification; or
    * Magnetic Resonance Angiography (MRA) confirming at least a 50% SFA or below the knee stenosis with moderate to severe calcification.
  * At least one patent, non-treated below the knee vessel.
  * Male and female patients that are ≥ 18 years of age.
  * Subject has been advised of the beneficial effects of smoking cessation and regular exercise but must not be in the process of changing their smoking status at the time of screening. Patients may resume or increase exercising as an effect of post procedurally improved lower limb perfusion.
  * Peak Walking Time (PWT) limited only by claudication.
  * Willingness to participate in the study, documented by signed, written informed consent.

Exclusion Criteria:

* • Planned amputation.

  * Any planned/scheduled revascularization procedures ≤ 30 days after baseline procedure.
  * Prior lower extremity revascularization ≤ 30 days before baseline procedure.
  * The target lesion is an in-stent restenosis.
  * Infra-popliteal disease involving the last remaining vessel.
  * Patients with a creatinine clearance < 30mL/min.
  * Patients with known bleeding disorders.
  * Patients with known active pathological bleeding.
  * Patients with known hypersensitivity to acetylsalicylic acid, clopidogrel bisulfate, ticagrelor, Aspirin, or other antiplatelets/anticoagulants.
  * Patients with known history of intracranial hemorrhage at any time, GI bleed in the past 6 months, or major surgery within the past 30 days.
  * Patients with known ischemic stroke during the past 3 months.
  * Patients with known severe liver disease.
  * Patient with known history of congestive heart failure (CHF) with an LVEF of < 30%.
  * Patients considered being at risk of bradycardic events unless treated with a permanent pacemaker.
  * Female patients with known pregnancy, breast feeding, or intend to become pregnant during the study period (all female patients 55 years and younger, without a history of hysterectomy must have a pregnancy test prior to PPI at baseline and at 6 months).
  * Concern for inability of the patient to comply with study procedures and/or follow up (e.g., alcohol or drug abuse).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2019-05-13 (Actual); Study Completion 2019-05-13 (Actual)

PRIMARY OUTCOMES:
Change in luminal area gain, measured in mm, in treated segment of the vessel wall | Baseline and 7 month
  Luminal area gain in the treated segment of the vessel wall between pre-and post-atherectomy OCT images.

SECONDARY OUTCOMES:
Atherectomy OCT Analysis-plaque volume | 0 and 7 months
  Changes in calcified total plaque volume as compare to baseline.
Atherectomy OCT Analysis-fibrous tissue | 0 and 7 months
  Changes in fibrous tissue amount as compared to baseline
Atherectomy OCT Analysis- new dissections | 0 and 7 months
  Number of new dissections present at 7 months as compare to baseline
Atherectomy OCT Analysis-new injuries | 0 and 7 months
  Percentage of cross-sectional images with new injury to the adventitia or EEL as compared to baseline
Atherectomy images Analysis-Luminal area loss | 0 and 7 months
  Change in Luminal area loss as measure by calcified plaque volume as well as by the presence of lipid and fibrous tissue as compared to baseline
Atherectomy images Analysis-persistent dissections | 0 and 7 months
  Percentage of cross-sectional images with persistent dissections as compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Cilingiroglu, MD, Principal Investigator — Arkansas Heart Hospital
Locations (2):
- United States (2):
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Arkansas Site Management Services LLC, Little Rock, Arkansas

IPD SHARING:
Plan to Share IPD: No